CLINICAL TRIAL: NCT01591265
Title: SIXES: Should I eXtract Every Six? A Randomized Clinical Trial of the Extraction of First Permanent Molar Teeth in Children
Brief Title: SIXES: Should I eXtract Every Six? A Study of the Extraction of Permanent Molar Teeth in Children.
Acronym: SIXES
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor recruitment
Sponsor: Professor David Bearn (Other)
Collaborators: NHS Tayside (Other Government)
Responsible Party: Sponsor-Investigator, Professor David Bearn, Cheif Investigator, University of Dundee
Organization: University of Dundee (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011DE02
Record Dates: First submitted 2012-04-30; First posted 2012-05-03 (Estimated); Last update posted 2018-06-29 (Actual); Status verified 2018-06

CONDITIONS: Paediatric Dentistry
Keywords: Compensatory dental extraction; Children 7-11 years old

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Compensatory Extraction (Active Comparator): Patients allocated to this group, both the upper FPM and lower FPM teeth will be extracted.
  Interventions: Procedure: Extraction of upper and lower FPM teeth
- No Compensatory Extraction (Active Comparator): Patients allocated to this group, only the lower FPM tooth will be extracted.
  Interventions: Procedure: Extraction of lower FPM tooth

INTERVENTIONS:
Procedure: Extraction of upper and lower FPM teeth — Extraction of upper and lower FPM teeth
  Arms: Compensatory Extraction
Procedure: Extraction of lower FPM tooth — Extraction of lower FPM tooth only
  Arms: No Compensatory Extraction

SUMMARY:
This clinical trial investigates relative benefits (clinical effectiveness and quality of life) of two extraction patterns when lower first permanent molars (FPM) are extracted in children The study objectives are to determine whether compensating extraction of upper FPMs following loss of lower FPMs in children is of benefit. The particular benefits being investigated are related to the resulting occlusion, patient experience and oral health related quality of life. The follow up will extend over a period of 5 years or until the patient is 14 years of age - whichever is earlier.

DETAILED DESCRIPTION:
The study has been designed as a randomised controlled clinical trial. The control group will have the normal standard intervention receiving routine patient care with the normal practice of upper and lower extractions, whilst the intervention group will have removal of the lower tooth but no upper extraction. Study recruitment will take place over an 18 month period and will be based in the Dundee Dental Hospital Orthodontic and Paediatric Dentistry Departments. Patients are referred to this department from their General Dental Practitioner.

Consent of the patients will be carried out by the attending dentists who will have received training on the study design and protocol, including RGF and consenting patients for clinical trials.

Data will be collected contemporaneously using the Case Report Forms. Additional data which will be collected for the purposes of the study will include COHQoL questionnaires and measurements from 3D images of models of the teeth.

At subsequent 1 year and five year review visits dental study 3D models will be repeated, and the CRF completed together with the COHQoL questionnaire for that visit.

ELIGIBILITY:
Inclusion Criteria:

* Age: 7 -11 years
* Dental History: Able to co-operate with dental treatment
* Regular attender or considered likely to return for follow-up Social History
* Child and carer able to understand study documentation and give consent to participate in study

Dental condition:

* One or two lower FPMs requiring extraction
* Upper FPMs are sound or restorable/ restored with good long term prognosis (i.e. has or requires a single surface restoration with caries less than half-way into dentine, restoration with a simple restoration)
* Confirmed presence of all second premolars and all second molars

Exclusion Criteria

* Medical History: Medical contraindication to dental extractions
* Dental condition: Poor prognosis of premolars or permanent second molar teeth
* All four upper incisors in crossbite
* Poor prognosis of upper FPM
* Confirmed absence of one or more second premolars and second molars
* Declines to have impressions taken

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 7 (Actual)
Dates: Start 2014-05; Primary Completion 2015-03-25 (Actual); Study Completion 2015-03-25 (Actual)

PRIMARY OUTCOMES:
Extent of tipping of the lower second permanent molars | 5 year
  The primary outcome measure is extent of tipping of the lower second permanent molar, with a favourable outcome being a degree of tipping less than 15°, and unfavourable outcome being greater than 15°.
  Participants will be allocated into 'favourable' or 'unfavourable' outcome groups when comparing study models, cast from dental impressions taken at baseline with 1 year and 5 year follow up or when the patient reaches 14 years of age, whichever is first.

SECONDARY OUTCOMES:
position of the upper FPMs with regard to over-eruption | 1 year and 5 year
  The secondary outcomes for the study are:
  1.position of the upper FPMs with regard to over-eruption;Outcome will be measured on study models of the teeth, cast from impressions taken at baseline and after 1 year and 5 years or when the participant reaches 14 years of age, whichever is first.
residual spacing between the lower second permanent molar and the lower second premolar*; | 1 year and 5 year
  Outcome be measured on study models of the teeth, cast from impressions taken at baseline and after 1 year and 5 years or when the participant reaches 14 years of age, whichever is first.
American Board of Orthodontics (ABO) scores | 1 year and 5 year
  Outcome will be measured on study models of the teeth, cast from impressions taken at baseline and after 1 year and 5 years or when the participant reaches 14 years of age, whichever is first.
the type of anaesthetic used during procedures | at baseline only
  Compare whether there is a difference in the type of anesthetic used by the dentist dependent on the intervention allocated.
dental or orthodontic treatment carried out during the follow-up period | 1 year and 5 year
  To compare if there is a difference in the frequency or type of dental or orthodontic treatment between the two groups of children.
Child and Parent Oral Health Related Quality of Life (OHRQoL) scores | 1 year and 5 year
  Child and Parent Oral Health Related Quality of Life (OHRQoL) scores (child and parent questionnaires)will be assessed at one year and 5 year follow up and compared with baseline.

CONTACTS AND LOCATIONS:
Overall Officials: David R Bearn, MOrth MFDS, Principal Investigator — University of Dundee; Nicola Innes, PhD, MFDS,, Principal Investigator — University of Dundee
Locations (5):
- United Kingdom (5):
  - Springfield Community Dental Practive, Arbroath, Angus
  - Dumfries & Galloway Royal Infirmary, Dumfries, Dumfries & Galloway
  - Dundee Dental School, University of Dundee, Dundee, Tayside
  - Kingscross Hospital Community Dental Service, Dundee, Tayside
  - Broxden Community Dental Practice, Perth, Tayside

REFERENCES:
- [Derived] Innes N, Borrie F, Bearn D, Evans D, Rauchhaus P, McSwiggan S, Page LF, Hogarth F. Should I eXtract Every Six dental trial (SIXES): study protocol for a randomized controlled trial. Trials. 2013 Feb 27;14:59. doi: 10.1186/1745-6215-14-59. PMID 23442547